CLINICAL TRIAL: NCT04996602
Title: Therapeutic Efficiency and Response to 2.0 GBq (55mCi) 177Lu-EB-PSMA in Patients With mCRPC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PekingUMCH Lu-EB-PSMA
Record Dates: First submitted 2021-07-22; First posted 2021-08-09 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2.0 GBq of 177Lu-EB-PSMA (Experimental): The patients were intravenously injected with the dose about 2.0 GBq (55 mCi) of 177Lu-EB-PSMA and underwent 68Ga-PSMA PET/CT scans before and after the treatment.
  Interventions: Drug: 2.0 GBq of 177Lu-EB-PSMA

INTERVENTIONS:
Drug: 2.0 GBq of 177Lu-EB-PSMA — Patients were intravenous administrated with the dose about 2.0 GBq (55 mCi) of 177Lu-EB-PSMA every 8 weeks (±1 week) for a maximum of 3 cycles.

SUMMARY:
In recent years, quite a few studies have demonstrated the possibility of 177Lu-PSMA-617 therapy as a viable treatment option in metastatic castration resistant prostate cancer (mCRPC), which has been shown desired effect. To increase tumor accumulation and retention for radioligand therapy, and reduce dosage of 177Lu, we conjugated a truncated Evans blue (EB) molecule and DOTA chelator onto PSMA-617 (EB-PSMA) and labeled it with 177Lu. This study is designed to assess the efficiency and response to 177Lu-EB-PSMA (55 mCi) in patients with mCRPC.

DETAILED DESCRIPTION:
Prostate cancer is one of the most common cancers and the second most frequent cause of cancer deaths for adult men. With the advances in the diagnosis and treatment of prostate cancer, some patients with localized prostate cancer can achieve good curative results, but there are still 10%～20% of patients progress to metastatic castration-resistant prostate cancer (mCRPC) every year, only one third of patients with mCRPC survive more than five years. Radioligand therapy targeting prostate specific membrane antigen (PSMA), which is overexpressed in most prostate cancer and even further increased in metastatic and castration-resistant carcinomas, has been demonstrated as an effective and safe therapy in men with mCRPC. 177Lu-PSMA-617 has also shown desired effect. However, 177Lu-PSMA-617, as a small molecule imaging agent, is cleared very quickly from the circulation. Therefore, radiotherapy that is based on small molecules requires high doses and frequent administrations, leading to systemic toxicity. To increase tumor accumulation and retention for radioligand therapy, and reduce dosage of 177Lu, the investigators conjugated a truncated Evans blue (EB) molecule and DOTA chelator onto PSMA-617 (EB-PSMA) and labeled it with 177Lu. The investigators have published some articles demonstrated 177Lu-EB-PSMA had much higher accumulation in prostate cancer lesions than 177Lu-PSMA-617 and also showed an ideal effect. This study is designed to assess the efficiency and response to 177Lu-EB-PSMA (55 mCi) in patients with mCRPC.

ELIGIBILITY:
Inclusion Criteria:

* All the patients had progressive metastatic castration-resistant prostate cancer that did not respond to androgen-suppression therapy and/or systemic chemotherapy;
* Distant metastases with high PSMA expression were confirmed on 68Ga-PSMA PET/CT within one week before the injection of 177Lu-EB-PSMA.

Exclusion Criteria:

* The exclusion criteria were a serum creatinine level of more than 150 μmol per liter, a hemoglobin level of less than 10.0 g/dl, a white-cell count of less than 4.0× 109/L, a platelet count of less than 100 × 109/L, a total bilirubin level of more than 3 times the upper limit of the normal range and a serum albumin level of more than 3.0 g per deciliter, cardiac insufficiency including carcinoid heart valve disease, a severe allergy or hypersensitivity to radiographic contrast material, claustrophobia.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic effect: PSA Response | through study completion, an average of 1 month
  The serum PSA response was documented monthly until 8 weeks after the last treatment therapy, which can effectively reflect the treatment effect of prostate cancer. Biochemical response was classified as the following: partial response (PR) if PSA decrease ≥50%, progressive disease (PD) if PSA increase ≥ 25% and stable disease (SD) if PSA increase <25% or PSA decrease <50%.
Therapeutic effect: 68Ga-PSMA PET/CT Response | through study completion, an average of 2 months
  68Ga-PSMA-617 wholebody PET/CT acquisitions 8 weeks after each cycle of treatment. The molecular response was classified according to adapted modified PERSIST 1.0 criteria. Complete response (CR) was complete resolution of 68Ga-PSMA-617 uptake in the target lesions. Partial response (PR) was defined as ≥30% decrease in the SUVmax of the target lesions and total Lesions PSMA from the baseline scan, and ≥ 30% increase in the SUVmax value of the target lesions and total Lesions PSMA from the baseline scan was taken as progressive disease (PD). Neither CR, PR nor PD was considered stable disease (SD) that was <30% decrease or <30% increase of the target lesion. Changes of SUV (ΔSUV) between pre- and post-therapeutic PET were calculated.

SECONDARY OUTCOMES:
Adverse events collection: Blood tests | through study completion, an average of 1 month
  Blood tests including hematologic status, liver function, and renal function were performed before and every two weeks after each cycle of treatment for a period of 8 weeks. Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China